CLINICAL TRIAL: NCT02761993
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Efficacy, and Treatment Regimen of ST266 in Subjects With Moderate to Severe Periodontitis
Brief Title: Safety, Efficacy and Treatment Regimen Study of ST266 in Subjects With Moderate to Severe Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST266-PERIO-201
Record Dates: First submitted 2016-04-21; First posted 2016-05-04 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Group 1 received ST266 treatment daily on Days 1 through 5, 8 through 12, 22, and 30, and then monthly for 7 months (Days 60, 90, 120, 150, 180, 210, and 240).
  Interventions: Biological: ST266
- Group 2 (Active Comparator): Group 2 received ST266 treatment 2x/week (with at least 1 day between treatments) for the first 3 months, and then monthly for 5 months (Days 120, 150, 180, 210, and 240).
  Interventions: Biological: ST266
- Group 3 (Placebo Comparator): Group 3 received commercially available sterile saline (0.9% sodium chloride) according to the same schedule as Group 1.
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Biological: ST266 — 1X ST266 applied in a dose of 20 microliters per tooth. Total daily dose will be less than 1 milliliter. ST266 will be applied directly to the marginal gingiva around each tooth (buccal and lingual).
  Arms: Group 1; Group 2
Drug: Saline (0.9% NaCl) — Saline applied in a dose of 20 microliters per tooth. Total daily dose will be less than 1 milliliter. Saline will be applied directly to the marginal gingiva around each tooth (buccal and lingual).
  Arms: Group 3

SUMMARY:
The purpose of this study is to determine whether ST266 will reduce pocket depth (PD) as an adjunctive to scaling and root planing (SRP) in subjects with moderate to severe periodontal disease.

DETAILED DESCRIPTION:
The study is a 9-month, randomized, double-blind, parallel-design study of subjects with existing moderate to severe periodontal disease randomly assigned to one of three groups. The primary endpoint of PD change will be evaluated following 9 months of treatment. Subjects will be followed for 9 months for safety and radiographic evaluations.

Subjects who meet inclusion criteria will be randomized to one of three treatment groups.

Randomization will be stratified by site and smoker status (never smoked or quit smoking more than two years ago vs. has smoked within the last two years). Randomization will be blocked such that assignment to treatment groups both within sites and within smoker status will be approximately even (1:1:1). Treatment will be initiated after SRP.

All subjects will be evaluated at baseline and Days 1, 15, 30, 60, 90, 180, and 270.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written informed consent prior to participation in any study-related procedures.
* Good general health as evidenced by medical history.
* Between 18 and 85 years of age at time of informed consent signature.
* Male or female.
* Minimum of 18 teeth, excluding third molars.
* Having moderate to severe periodontal disease according to AAP definition (at least 6 teeth ≥6 mm PD and ≥3 mm CAL at baseline).
* Having >30 percent bleeding sites upon probing.
* Willing to abstain from chewing gums and other mouth rinses for the study duration.
* Ability and willingness to attend all study visits and comply with all study visits and comply with all study procedures and requirements.
* Willingness to abstain from routine dental care.
* For women with reproductive potential, willingness to use highly effective contraception (e.g. licensed hormonal contraception, intrauterine device, abstinence, or vasectomy in partner).

Exclusion Criteria:

* Presence of orthodontic appliances.
* A soft or hard tissue tumor of the oral cavity.
* Any dental condition that requires immediate treatment, such as carious lesions.
* Participation in any other clinical study within 30 days of screening or during the study.
* Pregnancy or lactation. If a subject meets this criterion, she may be rescreened for study participation when she no longer meets this criterion.
* Antibiotic therapy within the last 30 days.
* Chronic use (≥3 times/week) of anti-inflammatory medications (e.g., non-steroidal anti inflammatory drugs, steroids). Low-dose aspirin (less than 325 mg daily) is allowed.
* Immunocompromised subjects.
* Subjects with cancer or a history of cancer within the last 5 years of screening.
* Any medical history or any concomitant medication that might affect the assessment of the study treatment or periodontal tissues, such as diabetes, nifedipine, phenytoin (Dilantin), or anticoagulant medications (e.g., warfarin [Coumadin] etc.).
* Involvement in the planning or conduct of the study.
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or interfere with interpretation of the subject's study results.
* Previous randomization for treatment in the present study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Alabama at Birmingham School of Dentistry, Birmingham, Alabama
  - Oral Health Research Institute, Indianapolis, Indiana
  - Forsyth Institute, Cambridge, Massachusetts
  - Columbia University College of Dental Medicine, New York, New York
  - Stony Brook School of Dental Medicine, Stony Brook, New York
  - University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 52 | 49 | 50
Completed | 50 | 43 | 46
Not Completed | 2 | 6 | 4
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 52 | 49 | 50 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.52) | 51.6 (11.91) | 52.5 (11.16) | 51.1 (11.88)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 55 years | 34 | 29 | 28 | 91
  55 - ≤ 65 years | 13 | 12 | 16 | 41
  > 65 years | 5 | 8 | 6 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 25 | 68
  Male | 30 | 28 | 25 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 9 | 35
  Not Hispanic or Latino | 39 | 36 | 40 | 115
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 14 | 15 | 38
  White | 25 | 23 | 22 | 70
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 13 | 10 | 7 | 30
Smoking Status [Count of Participants; unit: Participants] — A smoker was a subject who had smoked within the past 2 years. A nonsmoker was a subject who had never smoked or had quit smoking more than 2 years ago.
  Participants
    Smoker | 13 | 14 | 13 | 40
    Non-Smoker | 39 | 35 | 37 | 111

OUTCOME MEASURES:

1. Primary Outcome: Changes in Pocket Depth (PD) for Those Pockets ≥ 6 mm at Baseline
Description: The primary efficacy endpoint of this study is the change from baseline in the PD at 9 months (Day 270) for those pockets ≥6 mm at baseline.
Time Frame: Baseline; 9 months
Population: Intention-to-Treat (ITT) population: All randomized subjects with non-missing data for a given endpoint and time point. If the proportion of subjects (and oral sites) with missing data is ≤5 percent, as we expect it to be, for these analyses we will use the non-missing data and ignore the missingness.
Measure: Mean (Standard Deviation); unit: Pocket Depth (mm)
Units Other Than Participants: Tooth-Sites
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 52 | 49 | 50
Number analyzed (Tooth-Sites) | 1323 | 1338 | 1374
Pocket Depth (mm)
  Pocket Depth (mm) - Baseline | 6.6 (0.93) | 6.6 (1.02) | 6.7 (1.03)
  Pocket Depth (mm) - Day 270: number analyzed (Participants) | 50 | 45 | 46
  Pocket Depth (mm) - Day 270: number analyzed (Tooth-Sites) | 1286 | 1211 | 1249
  Pocket Depth (mm) - Day 270 | 4.5 (1.45) | 4.6 (1.53) | 4.5 (1.49)
  Pocket Depth (mm) - Change from Baseline: number analyzed (Participants) | 50 | 45 | 46
  Pocket Depth (mm) - Change from Baseline: number analyzed (Tooth-Sites) | 1286 | 1211 | 1249
  Pocket Depth (mm) - Change from Baseline | -2.1 (1.40) | -2.0 (1.39) | -2.1 (1.44)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Test type: Superiority; p = 0.341, Generalized Estimating Equation — Since there were two (2) primary hypotheses, Bonferroni corrections were used to control for multiplicity, with p < 0.025 considered significant; Generalized estimating equations (GEE) method with a linear link and exchangeable covariance matrix (with subject correlation structure)
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Test type: Superiority; p = 0.774, Generalized Estimating Equations — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Changes in Clinical Attachment Level (CAL)
Description: Change in Clinical Attachment Level (CAL) (the measurement of the position of the soft tissue in relation to the cemento-enamel junction (CEJ) that is a fixed point, using probing depth and the distance from the gingival margin to the CEJ.) from baseline in CAL at 9 months (Day 270) in tooth sites with baseline PD ≥ 6mm.
Time Frame: Baseline, 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Clinical Attachment Level (mm)
Units Other Than Participants: Tooth-Sites
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 52 | 49 | 50
Number analyzed (Tooth-Sites) | 1323 | 1338 | 1374
Clinical Attachment Level (mm)
  Clinical Attachment Level (mm) - Baseline | 6.7 (1.69) | 6.8 (1.62) | 6.7 (1.7)
  Clinical Attachment Level (mm) - Day 270: number analyzed (Participants) | 50 | 45 | 46
  Clinical Attachment Level (mm) - Day 270: number analyzed (Tooth-Sites) | 1287 | 1229 | 1251
  Clinical Attachment Level (mm) - Day 270 | 5.1 (2.01) | 5.1 (1.92) | 5.1 (2.05)
  Clinical Attachment Level (mm) - Difference from Baseline: number analyzed (Participants) | 50 | 45 | 46
  Clinical Attachment Level (mm) - Difference from Baseline: number analyzed (Tooth-Sites) | 1287 | 1229 | 1251
  Clinical Attachment Level (mm) - Difference from Baseline | -1.6 (1.48) | -1.7 (1.79) | -1.6 (1.60)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Test type: Superiority; p = 0.501, Generalized Estimating Equations — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Test type: Superiority; p = 0.486, Generalized Estimating Equations — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Bleeding on Probing (BOP)
Description: A secondary efficacy endpoint of this study is change from baseline in BOP at 9 months (Day 270) with BOP for each subject calculated as the percentage of tooth sites in the whole mouth with BOP.
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: Percentage of bleeding tooth-sites
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 52 | 49 | 50
Percentage of bleeding tooth-sites
  Bleeding on Probing (%) - Baseline | 67 (17.51) | 62.8 (15.84) | 67.5 (19.15)
  Bleeding on Probing (%) - Day 270 | 40.9 (20.80) | 38.8 (19.96) | 41.7 (25.2)
  Bleeding on Probing (%) - Change from Baseline | -26.2 (18.52) | -24.0 (21.23) | -25.8 (19.42)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Test type: Superiority; p = 0.816, ANCOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Test type: Superiority; p = 0.706, ANCOVA

ADVERSE EVENTS:
Time Frame: Events that occurred after first treatment dose date and prior to the last treatment dose date + 30 days, a total of up to 9 months
Groups:
- Group 1: Group 1: 1XST266 dosed as per regimen 1.
  ST266: 1X ST266 applied in a dose of 20 microliters per tooth. Total daily dose will be less than 1 milliliter. ST266 will be applied directly to the marginal gingiva around each tooth (buccal and lingual).
- Group 2: Group 2: 1XST266 as per regimen 2.
  ST266: 1X ST266 applied in a dose of 20 microliters per tooth. Total daily dose will be less than 1 milliliter. ST266 will be applied directly to the marginal gingiva around each tooth (buccal and lingual).
- Group 3: Group 3: Placebo dosed as per regimen 1.
  Saline (0.9% NaCl): Saline applied in a dose of 20 microliters per tooth. Total daily dose will be less than 1 milliliter. Saline will be applied directly to the marginal gingiva around each tooth (buccal and lingual).
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/52 | 2/49 | 2/50
Other Adverse Events (participants affected / at risk) | 29/52 | 27/49 | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=52) | Group 2 (N=49) | Group 3 (N=50)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=52) | Group 2 (N=49) | Group 3 (N=50)
Gingival pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gingival erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Leukoplakia oral (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4) | 1 (1)
Dental fistula (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Mouth injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
Burn oral cavity (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Tongue injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 7 (7) | 5 (5) | 3 (3)
Blood pressure systolic increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Device failure (Product Issues) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral mucosal exfoliation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Palatal swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth resorption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Traumatic occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gingival injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin urine (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Device damage (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT02761993/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT02761993/SAP_001.pdf